CLINICAL TRIAL: NCT00810173
Title: Phone Call as an Intervention for Improving Walking Practice in Type 2 Diabetes: Influence of Personality Profile in This Response
Brief Title: Phone Call in Type 2 Diabetes Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Cristina Helena Ferreira Fonseca-Guedes, Hospital das Clínicas da Universidade de São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Fonseca-Guedes
Record Dates: First submitted 2008-12-16; First posted 2008-12-17 (Estimated); Last update posted 2008-12-17 (Estimated); Status verified 2008-12

CONDITIONS: Behavior Change
Keywords: type 2 diabetes; physical activity; behavior change; profile personality; phone call support
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): This group received call phone support to incentive the increase of the number of steps during 6 weeks
  Interventions: Behavioral: phone call support
- 2 (No Intervention): This group just received a pedometer to register the number of steps for 6 weeks but this group don´t received a phone call.

INTERVENTIONS:
Behavioral: phone call support — The intervention group received a phone call support for 6 weeks to incentive to increase the number of steps/day.
  Other Names: couselling to behavior change
  Arms: 1

SUMMARY:
To assay the influence of personality profile to promote behavior change adherence for physical activity using a pedometer. The investigators also studied the metabolic profile, diagnosis of depression, intention to change behavior, physical activity referred and the quality of life. Casuistic and Methods: a randomized "quasi-experimental" enrolling 48 T2DM patients using a pedometer for 6 weeks. The intervention group received phone calls stimulating them to increase their walking activity. The control group received only one telephone call to explain pedometer use. The investigators also analyzed the personality profile, quality of life, and metabolic and anthropometric indexes.

ELIGIBILITY:
Inclusion Criteria:

* to assign written informed consent
* to have a phone call number
* to agree to use a pedometer for 6 weeks to be able to write the data concerning their number of steps per day

Exclusion Criteria:

* don´t agree to assign written informed consent
* don´t have phone number
* don´t have conditions to answer all the questionnaire
* don´t agree to use pedometer for 6 weeks

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2008-01; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)